CLINICAL TRIAL: NCT05830279
Title: Evaluating the Implementation of Personalized Medicine for Optimal Drug Therapy in Cancer Patients: A Prospective Longitudinal Trial
Brief Title: Implementation of Personalized Medicine for Optimal Drug Therapy in Cancer
Status: Recruiting | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Richard Kim, Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: 11642
Record Dates: First submitted 2023-04-13; First posted 2023-04-26 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Nausea With Vomiting Chemotherapy-Induced; Depression, Reactive; Cancer Pain
Keywords: Personalized medicine; Pharmacogenetics; Therapeutic drug monitoring
MeSH Terms: conditions — Adjustment Disorders; Cancer Pain | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be collected at each in-person appointment for extraction of DNA (genotype) and plasma (drug level analysis).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Anti-depressants: Patients who have been prescribed either 1) the selective serotonin reuptake inhibitors (SSRI) citalopram or escitalopram, or 2) the selective norepinephrine reuptake inhibitors (SNRI) venlafaxine or desvenlafaxine
  Interventions: Genetic: Pharmacogenetic testing; Other: Drug-Drug interaction analysis
- Opioid pain medications: Patients who have been prescribed opioid pain medications including codeine, oxycodone, hydrocodone, or tramadol.
  Interventions: Genetic: Pharmacogenetic testing; Other: Drug-Drug interaction analysis
- Anti-metics: Patients who have been prescribed the antiemetic agent ondansetron
  Interventions: Genetic: Pharmacogenetic testing; Other: Drug-Drug interaction analysis

INTERVENTIONS:
Genetic: Pharmacogenetic testing — Genotyping for CYP2D6 and CYP2C19
Other: Drug-Drug interaction analysis — Evaluating potential drug interactions with CYP2D6, CYP2C9 and CYP3A4 inhibitors and inducers using the Medical Letter.

SUMMARY:
A prospective longitudinal cohort study that will assess the effect of a Personalized Medicine (PM) clinic recommendations on pharmacogenetic variation and/or interacting drugs on plasma drug exposure, effectiveness or toxicity of commonly used antidepressant, pain, and antiemetic medications in cancer patients. Such recommendations will entail genotype-guided treatment suggestions while also considering potential DDI, and will be provided to patients during their clinic visit, and referring physicians thereafter. Drug concentration and therapeutic effectiveness will be assessed before (baseline) and 6 months after recommendations have been provided. To assess effectiveness, patient-reported outcomes will be evaluated using validated scales for symptoms of depression, pain and chemotherapy-induced nausea/ vomiting

The investigators hypothesize that the pharmacogenetic variation and DDI, if applicable, determine steady state drug concentration and therapeutic response or toxicity of the investigated antidepressant, pain or antiemetic treatments at baseline, while there is a clinically significant reduction or absence of the effect 6 months after the PM clinic recommendations to referring physicians and patients.

DETAILED DESCRIPTION:
This prospective longitudinal study will consist of three cohorts of adult cancer patients routinely referred to the PM clinic for genotype-guided chemotherapy including 5-FU or tamoxifen that are also taking antidepressant, analgesic and/or antiemetic medications.

Patients will be assigned to one or more cohorts, as appropriate, at the screening visit: Cohort 1 (n=200) if prescribed antidepressants including the selective serotonin reuptake inhibitors (SSRI) citalopram or escitalopram, or the selective norepinephrine reuptake inhibitors (SNRI) venlafaxine or desvenlafaxine; Cohort 2 (n=200) if prescribed opioid pain medications including codeine, oxycodone, hydrocodone, or tramadol; and/or Cohort 3 (N=200) if prescribed the antiemetic agent ondansetron.

Each patient will participate in a PM clinic screening visit. Eligible patients will attend three subsequent study visits at 0.5, 4 (virtual), and 7 months after screening. At each PM clinic visit, clinical information and a venous blood sample will be collected. Patients will also complete the ESAS survey and validated scores/ surveys to evaluate treatment effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Prescribed a chemotherapy medication
* Currently taking one or more study medications (citalopram, escitalopram, venlafaxine, desvenlafaxine, codeine, oxycodone, hydrocodone, tramadol or ondansetron)

Exclusion Criteria:

* Patients who are unable to complete study materials (surveys) with or without assistance, including non-English speaking patients
* Patients receiving palliative care
* Patients taking anti-depressants for reason other than depression or anxiety, i.e. hot flash (Only applies to antidepressant cohort)
* Patients with preexisting major depressive disorder prior to cancer diagnosis (Only applies to antidepressant cohort)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients taking selective medications for treatment of chemotherapy side effects, pain, depression and nausea.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Drug level measurements | Baseline visit to 6 months
  Steady-state drug plasma concentration of the antidepressant (Cohort 1), pain (Cohort 2) or antiemetic medication (Cohort 3) at follow-up visit 2 at 6 months compared to the baseline visit as assessed by single time points

SECONDARY OUTCOMES:
Edmonton Symptom Assessment Scale (ESAS) Survey | Baseline visit to 6 months
  Difference in ESAS survey results in each cohort at the follow up visits (3 and 6 months) compared to baseline visit. 10 questions, scale for each question between 0-9, higher score is associated with worse outcomes.
Center for Epidemiologic Studies Depression Scale (CES-D) Survey | Baseline visit to 6 months
  Difference in CES-D survey results in each cohort at the follow up visits (3 and 6 months) compared to baseline visit. 20 questions, scale for each question between 0-3, higher score is associated with worse outcomes.
Visual Analog Scale (VAS) for pain | Baseline visit to 6 months
  Difference in VAS Pain score in each cohort at the follow up visits (3 and 6 months) compared to baseline visit. Scale 0-100, higher score is associated with worse outcomes.
MASCC Antiemesis Tool (MAT) survey | Baseline visit to 6 months
  Difference in MAT survey results in each cohort at the follow up visits (3 and 6 months) compared to baseline visit
Antidepressant Side-Effect Checklist (ASEC) | Baseline visit to 6 months
  Difference in ASEC score in each cohort at the follow up visits (3 and 6 months) compared to baseline visit. 21 questions, scale for each question between 0-3, higher score is associated with worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kim, MD, Principal Investigator — Western University, Canada
Locations (1):
- Lawson Health Research Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No